CLINICAL TRIAL: NCT01175980
Title: A Phase 2 Study of Suberoylanilide Hydroxamic Acid (SAHA) in Subjects With Locally Advanced, Recurrent or Metastatic Adenoid Cystic Carcinoma (ACC)
Brief Title: Vorinostat in Treating Patients With Locally Advanced, Recurrent, or Metastatic Adenoid Cystic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02981; NCI-2012-02981 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-165; 8474 (Other: Wayne State University/Karmanos Cancer Institute); 8474 (Other: CTEP); P30CA022453 (NIH); U01CA132123 (NIH); U01CA062487 (NIH); U01CA062502 (NIH); U01CA062505 (NIH)
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Recurrent Oral Cavity Adenoid Cystic Carcinoma; Recurrent Salivary Gland Carcinoma; Salivary Gland Adenoid Cystic Carcinoma; Stage III Major Salivary Gland Cancer AJCC v7; Stage III Oral Cavity Adenoid Cystic Carcinoma AJCC v6 and v7; Stage IVA Major Salivary Gland Cancer AJCC v7; Stage IVA Oral Cavity Adenoid Cystic Carcinoma AJCC v6 and v7; Stage IVB Major Salivary Gland Cancer AJCC v7; Stage IVB Oral Cavity Adenoid Cystic Carcinoma AJCC v6 and v7; Stage IVC Major Salivary Gland Cancer AJCC v7; Stage IVC Oral Cavity Adenoid Cystic Carcinoma AJCC v6 and v7; Tongue Carcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms; Tongue Neoplasms | interventions — Vorinostat

ARMS (1):
- Treatment (vorinostat) (Experimental): Patients receive vorinostat PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Vorinostat

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase II trial studies how well vorinostat works in treating patients with adenoid cystic carcinoma that has come back (recurrent) or that has spread from where it started to nearby tissue or lymph nodes (locally advanced) or has spread to other places in the body (metastatic). Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy by means of response rate (based on Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria) of vorinostat in the treatment of patients with locally advanced, recurrent or metastatic adenoid cystic carcinoma (ACC).

SECONDARY OBJECTIVES:

I. To characterize the safety and tolerability of vorinostat in this patient population.

II. To assess the time to tumor response (TTR). III. To assess the response duration (RD). IV. To evaluate progression free survival (PFS). V. To assess overall survival (OS).

TERTIARY OBJECTIVES:

I. To assess the association between a metabolic response by positron emission tomography (PET)/computed tomography (CT) after one cycle of chemotherapy and subsequent best tumor response according to standard anatomic response evaluation criteria (RECIST).

II. To assess the association between a metabolic response by PET/CT after the first and second chemotherapy cycle and PFS.

III. To assess flow sort diploid, aneuploid, and tetraploid populations of tumor cells from formalin fixed, paraffin-embedded (FFPE) tissue blocks from patients who benefited from suberoylanilide hydroxamic acid (SAHA) therapy and from patients who did not demonstrate a durable benefit.

IV. Profile the genomes of each cell population using oligonucleotide comparative genomic hybridization (CGH) arrays.

V. Perform whole exome analysis of the sorted tumor population and matching germ line sample for each of the patients selected.

VI. To assess stable disease duration (SDD). VII. To assess the association between response to vorinostat treatment and RAD23 homolog B (HR23B) on tumor paraffin blocks.

VIII. Retrospectively compare volumetric density (viable tumor volume = VTV) with pre-determined RECIST of target lesions in cross sectioning imaging (CT/magnetic resonance [MR]) already obtained.

IX. Correlate VTV, RECIST and treatment response (partial response, stable disease, progressive disease and stable disease over 6 months).

OUTLINE:

Patients receive vorinostat orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up for 180 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed locally advanced, recurrent or metastatic adenoid cystic carcinoma
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm by chest x-ray, as >= 10 mm with CT scan, or >= 10 mm with calipers by clinical exam; all tumor measurements must be recorded in millimeters (or decimal fractions of centimeters)
* Patients must have locally advanced and/or recurrent and/or metastatic disease not amenable to potentially curative surgery or radiotherapy; any prior number of chemotherapy regimens is allowed; a minimum of at least 4 weeks since prior chemotherapy or radiation therapy should have elapsed, 6 weeks if the last regimen included carmustine (BCNU) or mitomycin C
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits (WNL)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN)
* Creatinine within normal institutional limits or
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of vorinostat will be determined following review of their case by the principal investigator
* No other diagnosis of malignancy unless non-melanoma skin cancer, carcinoma in situ of the cervix, or a malignancy diagnosed >= 5 years previously and currently with no evidence of disease; however - if the patient has had a previously diagnosed stage I/II malignancy of another type, consideration for recruitment may be made by the Cancer Therapy Evaluation Program (CTEP) senior investigator after discussion with local principal investigator (PI) and patient's physician
* Confirmed availability of tumor tissue (either fresh or from paraffin block) from the primary tumor or metastatic site to be available to use on correlative studies
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* If the patient's tumor can be easily accessed, a pre-treatment biopsy will be mandatory

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; more than 21 days from major surgery should have elapsed before the first dose of the study drug
* Patients may not be receiving any other investigational agents or have received vorinostat in the past; patients should not have taken valproic acid for at least 4 weeks prior to enrollment
* Inability to take oral medications on a continuous basis
* Patients with active brain metastases should be excluded from this clinical trial; patients with previous brain metastases will be eligible if condition is treated and stable for >= 1 month
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SAHA
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with vorinostat
* Patient is unable or unwilling to abide by the study protocol and to cooperate fully with the investigator or designee
* Patient on current therapy with enzyme-inducing anticonvulsants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08-06 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia LoRusso, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (12):
- United States (11):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope South Pasadena, South Pasadena, California
  - Yale University, New Haven, Connecticut
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Veterans Administration, Cleveland, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Ireland Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Vorinostat)
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 53 [21 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 3
  Caucasian | 24
  Middle Eastern | 1
  Asian | 2
Region of Enrollment [Number; unit: participants]
  Canada | 5
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Objective Response According to RECIST 1.1 Criteria
Description: Objective (Best) response according to RECIST 1.1 criteria.
Time Frame: Up to 180 days after the last dose of vorinostat maximum treatment duration= 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 30
Participants
  Partial Response | 2
  Stable Disease | 27
  Progressive Disease | 1

2. Secondary Outcome: Number of Participants With Grade 3 or Grade 4 Toxicity as Assessed by the Common Terminology Criteria for Adverse Events Version 4.0
Description: Toxicity will be tabulated via frequency distributions, and also dichotomized to report the proportion (and percentage) of patients experiencing a specified level (e.g., grade 3-4) of toxicity.
Time Frame: Up to 180 days after the last dose of vorinostat maximum treatment duration= 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 30
Participants
  Appendicitis | 1
  Atelectasis | 1
  Bronchial obstruction | 1
  Bronchopulmonary hemorrhage | 1
  Cataract | 1
  Diarrhea | 1
  Fatigue | 3
  Headache | 2
  Hypertension | 3
  Hypophosphatemia | 1
  Hypoxia | 1
  Lung infection | 1
  Lymphocyte count decreased | 7
  Lymphocyte count increased | 1
  Menorrhagia | 1
  Mucositis oral | 1
  Non cardiac chest pain | 1
  Oral pain | 2
  Platelet count decreased | 1
  PNEUMONIA | 1
  Thromboembolic event | 2
  Wound complication | 1

3. Secondary Outcome: Time to Recurrence (TTR)
Description: TTR will be summarized descriptively, reporting N, median, mean, standard deviation, standard error (SE), minimum, maximum, and 90% CI for the mean calculated from the SE and asymptotic normal distribution theory.
Time Frame: From the start of the treatment until the RECIST measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded, assessed up to 180 days after the last dose of vorinostat maximum treatment duration= 24 months
Population: Only 2 patients achieved a response.
Measure: Mean (90% Confidence Interval); unit: months
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 2
months | 8.85 [1.59 to 16.11]

4. Secondary Outcome: Response Duration (RD)
Description: Median point estimate and full range will be documented, since only two patients achieved a response.
Time Frame: From the time measurement criteria are met for CR or PR (whichever is first) until the first date that recurrence or progression is objectively documented, assessed up to 60 months after the last dose of vorinostat max. treatment duration= 24 months
Population: Only 2 patients achieved a response.
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 2
months | 30.1 [7.2 to 53.0]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Distribution will be estimated using standard survival analysis techniques, and the K-M method. From the K-M life tables, both median point estimate and 90% confidence interval (CI) estimate.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 60 months after the last dose of vorinostat maximum treatment duration= 24 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 30
months | 11.4 [7.1 to 20.5]

6. Secondary Outcome: Overall Survival (OS)
Description: Distribution will be estimated using standard survival analysis techniques, and the K-M method. From the K-M life tables, both point and 90% CI estimates of various statistics of interest can be calculated (e.g., median, 6-month event-free rate, 12-month event-free rate, etc.). Statistical graphs of each K-M curve (with 90% CI lines) will be generated for visual display.
  (One year survival rate will be given since OS median was not reached due to too few events)
Time Frame: From the start of treatment until death from any cause, duration for reported probability= 1 year; survival data collected for up to a total of 60 months
Measure: Number (90% Confidence Interval); unit: percentage of participants surviving 1yr
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 30
percentage of participants surviving 1yr | 88 [75 to 100]

7. Other Pre Specified Outcome: Metabolic Response by PET/CT Scan
Description: Will assess the association between a metabolic response by PET/CT after one course of chemotherapy and subsequent best tumor response according to standard anatomic response evaluation criteria. Will also assess the association between a metabolic response by PET/CT after the first and second chemotherapy courses and PFS.
Time Frame: Up to 56 days
Population: We did not have funding to incorporate other imaging modalities, (such as PET/CT), or to utilize other measurement criteria (such as volumetric assessment). Therefore, these data were not collected
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Number of Patients With Flow Sort Diploid Populations of Tumor Cells From FFPE Tissue Blocks
Description: Number of patients with Flow sort diploid populations of tumor cells from FFPE tissue blocks reported as a count of participants.
Time Frame: Up to 180 days after the last dose of vorinostat maximum treatment duration= 24 months
Population: the two cases that had FFPE blocks for the study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 2
Participants | 2

9. Other Pre Specified Outcome: Number of Patients With Flow Sort Aneuploid Populations of Tumor Cells From FFPE Tissue
Description: Number of patients with Flow sort aneuploid populations of tumor cells from FFPE tissue. Reported as descriptive results.
Time Frame: Up to 180 days after the last dose of vorinostat maximum treatment duration= 24 months
Population: The two cases that had FFPE blocks for the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 2
Participants | 0

10. Other Pre Specified Outcome: Number of Patients With Flow Sort Tetraploid Populations of Tumor Cells From FFPE Tissue
Description: Number of patients with Flow sort tetraploid populations of tumor cells from FFPE tissue. Reported as descriptive results.
Time Frame: Up to 180 days after the last dose of vorinostat maximum treatment duration= 24 months
Population: The two cases that had FFPE blocks for the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 2
Participants | 2

11. Other Pre Specified Outcome: Unique Probes on the Oligonucleotide CGH Array as a Measure of the Genomic Profile of Each Cell Population.
Description: Genomic profile of each cell population using oligonucleotide CGH arrays. Reported as unique probes on the CGH array.
Time Frame: Up to 180 days after the last dose of vorinostat maximum treatment duration= 24 months
Population: One of the cases that had FFPE blocks for the study.
Measure: Number; unit: unique probes on the CGH arrays
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 1
unique probes on the CGH arrays | 442,892

12. Other Pre Specified Outcome: The Number of Genes Sequenced in the WES Assay as a Measure of the Whole Exome Profile of the Sorted Tumor Population and Matching Germ Line Sample
Description: Reported as descriptive results. The combined CGH array and exome data will be mined to identify genes and pathways that are targeted by select somatic events in each of the patient subsets.
Time Frame: Up to 180 days after the last dose of vorinostat maximum treatment duration= 24 months
Population: One of the cases that had FFPE blocks for the study.
Measure: Number; unit: Genes sequenced in the WES assay.
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 1
Genes sequenced in the WES assay. | 21,522

13. Other Pre Specified Outcome: Stable Disease Duration (SDD)
Description: SDD will be reported as descriptive results as a median point estimate and a 90% confidence interval (CI) estimate.
Time Frame: Up to 180 days after the last dose of vorinostat maximum treatment duration= 24 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 30
months | 11.4 [7.1 to 20.5]

14. Other Pre Specified Outcome: Expression Level of HR23B
Description: Exact logistic modeling investigation would yield a point and 90% CI estimate of the odds ratio for response.
Time Frame: Up to 180 days after the last dose of vorinostat maximum treatment duration= 24 months
Population: HR23B was not measured in any participant.
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the start of treatment until death from any cause, assessed up to 180 days after the last dose of vorinostat] maximum treatment duration= 24 months
Arm/Group | Treatment (Vorinostat)
All-Cause Mortality (participants affected / at risk) | 3/30
Serious Adverse Events (participants affected / at risk) | 20/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vorinostat) (N=30)
Appendicitis (Gastrointestinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cataract (Eye disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (7)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
Hypoxia (General disorders) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (2)
Lung infection (Infections and infestations) | 1 (3)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 8 (18)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Mucositis oral (General disorders) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral pain (General disorders) | 2 (2)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
Thromboembolic event (Blood and lymphatic system disorders) | 2 (2)
Wound complication (General disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vorinostat) (N=30)
Abdominal pain (General disorders) | 9 (24)
Abducens nerve disorder (Nervous system disorders) | 1 (22)
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 3 (5)
Acute kidney injury (Renal and urinary disorders) | 1 (3)
Alanine aminotransferase increased (Hepatobiliary disorders) | 11 (41)
Alkaline phosphatase increased (Hepatobiliary disorders) | 7 (44)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (General disorders) | 17 (131)
Amnesia (Nervous system disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (7)
Anemia (Blood and lymphatic system disorders) | 15 (52)
Anorexia (Metabolism and nutrition disorders) | 17 (145)
Anxiety (Nervous system disorders) | 3 (16)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 10 (33)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (18)
Bloating (Gastrointestinal disorders) | 4 (4)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (2)
Blood bilirubin increased (Blood and lymphatic system disorders) | 8 (24)
Blurred vision (Eye disorders) | 4 (16)
Bronchial infection (Infections and infestations) | 3 (3)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 2 (4)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Buttock pain (General disorders) | 1 (1)
Cheilitis (Skin and subcutaneous tissue disorders) | 1 (2)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Chills (General disorders) | 5 (5)
Chronic kidney disease (Renal and urinary disorders) | 1 (2)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (45)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (9)
CPK increased (Blood and lymphatic system disorders) | 1 (3)
Creatinine increased (Renal and urinary disorders) | 18 (132)
Dehydration (General disorders) | 6 (18)
Depression (Psychiatric disorders) | 2 (5)
Diarrhea (Gastrointestinal disorders) | 13 (40)
Dizziness (Ear and labyrinth disorders) | 4 (13)
Dry eye (Eye disorders) | 2 (4)
Dry mouth (General disorders) | 5 (28)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (9)
Dysgeusia (General disorders) | 10 (87)
Dyspepsia (Gastrointestinal disorders) | 1 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (22)
CERUMEN IMPACTION OF THE RIGHT EAR (Ear and labyrinth disorders) | 1 (1)
LEFT EAR CERUMEN (Ear and labyrinth disorders) | 1 (1)
Edema limbs (Vascular disorders) | 2 (9)
Epistaxis (Blood and lymphatic system disorders) | 2 (13)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (2)
DOUBLE VISION (Eye disorders) | 1 (7)
REDDENED SCLERA POST OUTSIDE PROCEDURE (Eye disorders) | 1 (1)
STYLE LOWER RIGHT EYELID (Eye disorders) | 1 (3)
Eye infection (Infections and infestations) | 1 (1)
Eye pain (Eye disorders) | 1 (6)
Eyelid function disorder (Eye disorders) | 1 (5)
Facial pain (General disorders) | 1 (2)
Fall (General disorders) | 1 (2)
Fatigue (General disorders) | 21 (202)
Fever (General disorders) | 1 (4)
Flank pain (General disorders) | 2 (6)
Flatulence (Gastrointestinal disorders) | 3 (4)
Floaters (Eye disorders) | 1 (2)
Flu like symptoms (General disorders) | 3 (7)
Flushing (General disorders) | 1 (2)
Gait disturbance (General disorders) | 2 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (8)
CHEWING FATIGUE (Gastrointestinal disorders) | 1 (2)
BELCHING (Gastrointestinal disorders) | 1 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (6)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (2)
Headache (General disorders) | 7 (14)
Hearing impaired (Ear and labyrinth disorders) | 1 (12)
Hematoma (Vascular disorders) | 1 (3)
Hemoglobinuria (Renal and urinary disorders) | 3 (8)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (3)
Hyperglycemia (Blood and lymphatic system disorders) | 2 (8)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (4)
Hyperkalemia (Blood and lymphatic system disorders) | 3 (5)
Hypermagnesemia (Renal and urinary disorders) | 11 (42)
Hypertension (Vascular disorders) | 13 (73)
Hypoalbuminemia (Hepatobiliary disorders) | 8 (34)
Hypocalcemia (Blood and lymphatic system disorders) | 2 (2)
Hypoglycemia (Blood and lymphatic system disorders) | 2 (3)
Hypokalemia (Blood and lymphatic system disorders) | 3 (6)
Hypomagnesemia (Blood and lymphatic system disorders) | 5 (5)
Hyponatremia (Blood and lymphatic system disorders) | 5 (24)
Hypophosphatemia (Blood and lymphatic system disorders) | 5 (12)
Hypotension (Vascular disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 3 (14)
VIRAL INFECTION (Infections and infestations) | 1 (1)
KNEE INJURY (Injury, poisoning and procedural complications) | 1 (3)
BACK INJURY (Injury, poisoning and procedural complications) | 1 (2)
Insomnia (General disorders) | 5 (11)
LDH ELEVATED (Investigations) | 5 (12)
ELEVATED BUN (Investigations) | 1 (9)
CREATININE KINASE INCREASED (Investigations) | 1 (2)
Irregular menstruation (Reproductive system and breast disorders) | 2 (12)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (11)
Localized edema (Vascular disorders) | 1 (4)
Lung infection (Infections and infestations) | 3 (4)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 16 (87)
Malaise (General disorders) | 1 (10)
Memory impairment (Nervous system disorders) | 1 (5)
Menorrhagia (Reproductive system and breast disorders) | 2 (3)
DECREASE IN SERUM PROTEIN (Metabolism and nutrition disorders) | 1 (6)
Mucositis oral (Gastrointestinal disorders) | 5 (12)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (39)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 5 (68)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Nausea (General disorders) | 18 (78)
Neck pain (General disorders) | 1 (3)
BENIGN OVARIAN CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Neuralgia (Nervous system disorders) | 1 (5)
Neutrophil count decreased (Blood and lymphatic system disorders) | 8 (26)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 3 (11)
Oculomotor nerve disorder (Nervous system disorders) | 1 (22)
Olfactory nerve disorder (Nervous system disorders) | 1 (21)
Oral pain (General disorders) | 1 (3)
Otitis media (Ear and labyrinth disorders) | 2 (10)
Pain (General disorders) | 1 (1)
Pain in extremity (General disorders) | 5 (37)
Palpitations (Cardiac disorders) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (2)
Paronychia (Infections and infestations) | 1 (1)
Pelvic pain (General disorders) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (21)
Personality change (Psychiatric disorders) | 1 (17)
Photophobia (Psychiatric disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 22 (155)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Infections and infestations) | 1 (1)
Postnasal drip (General disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (13)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
DECREASED EGFR (Renal and urinary disorders) | 1 (1)
STENT REMOVAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HIGHTENED SENSE OF SMELL (Respiratory, thoracic and mediastinal disorders) | 1 (3)
GROUND GLASS APPERANCE (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Sinus bradycardia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Infections and infestations) | 3 (14)
HAND - FOOT SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1)
MULTIPLE BUMPS ON HEAD (Skin and subcutaneous tissue disorders) | 1 (1)
BRITTLE NAILS (Skin and subcutaneous tissue disorders) | 1 (6)
SKIN PEELING ON HANDS (Skin and subcutaneous tissue disorders) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (3)
Skin infection (Infections and infestations) | 3 (3)
Somnolence (General disorders) | 1 (1)
Sore throat (General disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (2)
TOOTH EXTRACTION (Surgical and medical procedures) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (6)
Thromboembolic event (Vascular disorders) | 2 (16)
Tooth infection (Infections and infestations) | 1 (1)
Tremor (Nervous system disorders) | 1 (4)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 6 (13)
Urinary frequency (Renal and urinary disorders) | 1 (4)
Urinary tract infection (Infections and infestations) | 2 (4)
Vaginal infection (Infections and infestations) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 8 (14)
Watering eyes (Eye disorders) | 1 (1)
Weight gain (Metabolism and nutrition disorders) | 2 (4)
Weight loss (Metabolism and nutrition disorders) | 13 (65)
White blood cell decreased (Blood and lymphatic system disorders) | 13 (78)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT01175980/Prot_SAP_000.pdf